CLINICAL TRIAL: NCT06560554
Title: Evaluating the Effects of a Fermented Diet on Microbiome Diversity in Individuals With Long COVID
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lioudmila Karnatovskaia, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-005170
Record Dates: First submitted 2024-08-09; First posted 2024-08-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Long COVID
Keywords: Long COVID; anxiety; depression; gut microbiome; fermented foods
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Anxiety Disorders; Depression | interventions — Fermented Foods

STUDY DESIGN:
Intervention Model Description: Single center, longitudinal, randomized trial
Who Masked: Participant
Masking Description: Participants who are randomized to the control group will not be given information on increasing fermented foods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The subjects in the control arm will only complete the baseline and week 13 visits. They will not be asked to make any changes to their diet, only to document their regular diet 3 days a week.
  Interventions: Other: Control
- Treatment (Experimental): Will receive an in-person teaching session delivered by a trained team member including introductory education on microbiome and a description on a variety of probiotic fermented foods commercially available (fermented dairy products, fermented vegetables, fermented non-alcoholic drinks). Participants will be able to choose their own probiotic fermented foods based on this education and taste preference. Subjects will be contacted weekly to ensure they are tolerating and adhering to the study protocol.
  Interventions: Other: Fermented foods

INTERVENTIONS:
Other: Fermented foods — Participants randomized to the intervention arm will begin to incorporate probiotic fermented foods into their diet during weeks 1-4 of the study (ramp up phase). They will start with one serving of fermented food of their choice a day, increasing to 6+/day as tolerated by the end of week 4. Weeks 5-12 will serve as the intervention maintenance phase, with the target of a daily intake of 6+ servings of fermented foods.
  Arms: Treatment
Other: Control — No information on incorporation of fermented foods will be provided for subjects in the control arm.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of fermented foods on bacterial gut microbiome diversity of long-COVID subjects.

DETAILED DESCRIPTION:
This will be a single-center, longitudinal randomized controlled trial assessing a high fermented food diet intervention among patients with long COVID.

The investigators will adapt the high fermented food diet intervention previously described by Wastyk et al to our population of patients with long COVID. A list of people meeting inclusion criteria who are open to research participation will be generated by the study team members working in the long COVID clinic; eligible patients will be contacted by a different member of the study team (not working in the long COVID clinic).

Participants who agree to take part in the study will be randomized using REDCap into one of two arms, a control arm (no diet intervention), or an intervention arm. 20 participants will be assigned to each group (40 total). The study will consist of 2 in-person visits at baseline and week 13. There will be weekly phone calls during weeks 1 through 12 for participants on the intervention arm; participants in the control arm will be contacted as needed to ensure that they continue to document their diet three days a week.

All participants will provide a total of two stool samples (baseline and week 13), and undergo psychometric evaluation with Hospital Anxiety and Depression Scale (HADS) A/D, Impact of Event Scale - revised (IES-R), Montreal Cognitive Assessment (MoCA)-blind and European Quality of Life 5 Dimensions 5 Level Version (EuroQol-5D-5L) (baseline and week 13). Demographic information on the subjects will also be collected (age, gender, past medical history including mental health diagnoses or cognitive diagnoses, time of COVID infection, etc).

During the baseline visit, the investigators will interview all study participants and ask participants to provide details about their diet and any use of probiotic foods or supplements. All participants will install the food tracking application, Mayo Clinic Diet App, on their personal smart device and will receive instructions on how to use it by a study team member. An account for each participant will be set up by the study team and participants will be given a username and password. The investigators will have access to the data entered. Participants will be instructed to document their food intake at least three days every week, two weekdays and one weekend day as was done in the study by Wastyk et al. After the study, participants may change their password if they would like to continue food tracking.

Intervention Group:

Participants assigned to the intervention arm will receive an in-person teaching session delivered by a trained team member. The session will include introductory education on microbiome and a description on a variety of probiotic fermented foods commercially available (fermented dairy products, fermented vegetables, fermented non-alcoholic drinks). Participants will be able to choose their own probiotic fermented foods based on this education and taste preference.

After the visit, intervention arm participants will begin to incorporate probiotic fermented foods into their diet during weeks 1-4 of the study (ramp up phase). Participants will start with one serving of fermented food of their choice a day, increasing to 6+/day as tolerated by the end of week 4. Weeks 5-12 will serve as the intervention maintenance phase, with the target of a daily intake of 6+ servings per day of fermented foods.

Fermented food intake will be reported as the average number of servings per day for each week of the intervention. One serving of probiotic fermented foods will be defined as: kombucha, yogurt, kefir, buttermilk, kvass, other probiotic fermented liquids = 6 oz, kimchi, sauerkraut, other probiotic fermented veggies = 1/4 cup, vegetable brine drink/gut shot from approved list = 2 oz.

Food logs will be reviewed by the investigators to assess compliance and provide recommendations to increase amounts or variety of fermented foods in the diet as tolerated. Investigators will interact weekly with participants in the intervention arm by phone or zoom to review probiotic fermented food intake, answer questions, inquire about any gastrointestinal symptoms such as bloating or upset stomach, and provide motivation to continue with the diet. Study participants in the intervention arm will also be asked to assess their overall compliance with the diet on a scale of 0-10, with zero being "not at all" and 10 being "exactly as recommended [during the specific phase of the study]".

Control Group:

The participants in the control arm will only complete the baseline and week 13 visits. Participants in the control arm will be contacted as needed to ensure that they document their regular food intake 3 days a week. Control group participants will not be asked to make any changes to their diet, only to document their regular diet 3 days a week.

At approximately 13 weeks, all participants will collect and return a stool sample and repeat the study questionnaires. Participants will be able to complete the questionnaires in person, virtually, or by phone.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (> 18 years old)
2. Patients who have long COVID symptoms

   a. Long COVID will be defined as: i. A previously documented COVID + infection within the last year ii. A presence of neurological symptoms that started within 4 weeks of the COVID infection (fatigue, difficulty concentrating, depression, anxiety) as per CDC definition of Long Covid.
3. Own a smart device capable of downloading a food logging application. Able to understand and document informed consent
4. Seen in the Mayo Clinic long-COVID Clinic within the Department of General Internal Medicine

Exclusion Criteria:

1. History of dementia, moderate or severe cognitive dysfunction, developmental delay, psychotic disorders such as schizophrenia
2. Unable to tolerate oral foods
3. Potential contraindications to a fermented food diet (chronically immunosuppressed including organ transplant recipients)
4. Neutropenic as listed in the "active problems" list in the EMR
5. Undergoing chemotherapy at the time of consent
6. Taking MAOIs at the time of consent.
7. Active uncontrolled inflammatory bowel disease including ulcerative colitis, Crohn's disease, indeterminate colitis, irritable bowel syndrome (moderate or severe), infectious gastroenteritis, colitis or gastritis, Clostridium difficile infection (recurrent), malabsorptive diseases (such as Celiac disease), major surgery of the GI tract with the exception of cholecystectomy and/or appendectomy in the past 5 years, or any major bowel resection at any time.
8. A reported consumption of 2 servings of probiotic fermented food per day in their normal baseline diet.
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome diversity | At enrollment and completion of study (12 weeks)
  High-dimensional microbiome data representing taxonomic features of the microbiomes will be analyzed to decode the community structure and key components that are associated with the condition of interest

SECONDARY OUTCOMES:
Symptoms of depression and anxiety | At enrollment and completion of study (12 weeks)
  Measured using the self-reported Hospital Anxiety and Depression Scale (HADS). Total questions: 14. Anxiety 7, Depression 7. Each item is rated on a 4-point scale from 0 "absence" to 3 "extreme presence". Total score is 21 per subscale: 0 - 7: Normal levels of anxiety/depression; 8-10: Borderline abnormal; > 11: Abnormal
Assessment of cognition | At enrollment and completion of study (12 weeks)
  Measured using the Montreal Cognitive Assessment (MoCA-BLIND). Total questions:13. Memory 3 Attention 4 Language 3 Abstraction 2 Orientation 1. Subscores for each of the 5 sections are calculated. The total score is summed from the subscores, with a maximum score of 22. A score equal > 18 is considered normal cognition
Assessment of quality of life | At enrollment and completion of study (12 weeks)
  Measured using the self-reported EuroQol-5D-3L questionnaire. Total questions: 6. Mobility: 1, Self-Care: 1, Usual Activities: 1, Pain/discomfort: 1, Anxiety/depression: 1, Health State - Visual Analog Scale: 1. 3L - 3 levels of severity: no problems, some problems, extreme problems. The visual analog scale ranges from 0 to 100 with higher scores reflecting better perceived current health-related quality of life state.
Assessment of post-traumatic stress (PTSD) symptoms | At enrollment and completion of the study (12 weeks)
  Measured using Impact of Events-revised (IES-r). Total questions: 22. Intrusion 7, Avoidance 8, Hyperarousal 7. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Total scores are summed with higher scores indicating greater distress with regards to a specific event.

OTHER OUTCOMES:
Research participant's subjective assessment of study adherence | At enrollment and weekly, through completion of the study (12 weeks)
  During weekly phone calls, research participants will be asked to rate their adherence to the study protocol on a scale of 0 to 10, with zero being "not at all" and 10 being "exactly as recommended [during the specific phase of the study]".

CONTACTS AND LOCATIONS:
Overall Officials: Liousmila V Karnatovskaia, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wastyk HC, Fragiadakis GK, Perelman D, Dahan D, Merrill BD, Yu FB, Topf M, Gonzalez CG, Van Treuren W, Han S, Robinson JL, Elias JE, Sonnenburg ED, Gardner CD, Sonnenburg JL. Gut-microbiota-targeted diets modulate human immune status. Cell. 2021 Aug 5;184(16):4137-4153.e14. doi: 10.1016/j.cell.2021.06.019. Epub 2021 Jul 12. PMID 34256014